CLINICAL TRIAL: NCT00806065
Title: A Phase 1 Study of ENMD-2076 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of ENMD-2076 in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2076-CL-002
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ENMD 2076

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENMD-2076 (Experimental): Oral capsules, once daily in 28-day cycles
  Interventions: Drug: ENMD-2076

INTERVENTIONS:
Drug: ENMD-2076

SUMMARY:
Safety, tolerability, maximum tolerated dose and clinical benefit of ENMD-2076 administered over a range of doses in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
The study is designed to assess the safety, tolerability, maximum tolerated dose, and clinical benefit of treatment with ENMD-2076 administered orally once daily over a range of doses in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Major Inclusion Criteria:

1. Histological evidence of MM and evidence of relapse or refractory disease. Patients with non secretory myeloma or plasmacytoma only will be excluded.
2. Patients must have failed thalidomide, lenalidomide, or velcade or be intolerant or ineligible to receive these agents.
3. Age ≥18 years.
4. ECOG performance status 0-2.
5. Patients must have adequate organ and marrow function

Major Exclusion Criteria:

1. Prior cytotoxic chemotherapy or investigational agent within 28 days or autologous stem cell transplant within 6 months of receiving study drug ENMD-2076.
2. Prior radiation therapy to > 25% of bone marrow forming bones (i.e., pelvis).
3. Concomitant corticosteroid therapy in doses greater than 10 mg daily of prednisone (or equivalent) if given for management of co-morbid conditions.
4. Have unstable angina pectoris or recent myocardial infarction (within 6 months.
5. Have uncontrolled hypertension or congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ENMD-2076 | Within first 35 days

SECONDARY OUTCOMES:
Correlative studies of activity | throughout the study period
Clinical Benefit | Each cycle of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No